CLINICAL TRIAL: NCT07395388
Title: Intraoperative Methylene Blue Spray for the Identification and Preservation of Vital Structures in Thyroidectomy: A Randomized Controlled Trial
Brief Title: Intraoperative Methylene Blue Spray for the Identification and Preservation of Vital Structures in Thyroidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Services Hospital, Lahore (Other Government)
Responsible Party: Principal Investigator, Dr. SamiUllah, Doctor, Services Hospital, Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RCT22SIMS
Record Dates: First submitted 2026-02-01; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Benign Multinodular Goiter; Thyroidectomy; Recurrent Laryngeal Nerve Injury; Hypoparathyroidism
Keywords: Thyroidectomy; Methylene Blue; Recurrent Laryngeal Nerve Injury; Hypocalcemia; Nerve Preservation
MeSH Terms: conditions — Recurrent Laryngeal Nerve Injuries; Hypoparathyroidism; Hypocalcemia

STUDY DESIGN:
Intervention Model Description: Experimental Group: Intraoperative topical spray of 0.5 mL methylene blue applied to the thyroid lobe and surrounding tissue after mobilization.
  Control Group: Conventional visual identification and dissection without dye.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methylene Blue labelling (Experimental)
  Interventions: Procedure: Intraoperative topical methylene blue spray
- Conventional Dissection (Active Comparator)
  Interventions: Procedure: Conventional Dissection

INTERVENTIONS:
Procedure: Intraoperative topical methylene blue spray — Intraoperative topical spray of 0.5 mL methylene blue applied to the thyroid lobe and surrounding tissue after mobilization.
  Arms: Methylene Blue labelling
Procedure: Conventional Dissection — Conventional visual identification and dissection without dye.
  Arms: Conventional Dissection

SUMMARY:
This randomized controlled trial aims to evaluate the efficacy of intraoperative methylene blue (MB) spray in improving the identification and preservation of the recurrent laryngeal nerve (RLN) and parathyroid glands (PGs) during thyroidectomy. The study compares outcomes between patients receiving topical MB spray and those undergoing conventional visual dissection alone. Primary outcomes include the incidence of RLN injury and postoperative serum calcium levels.

DETAILED DESCRIPTION:
Thyroidectomy is associated with risks of iatrogenic injury to the RLN and PGs, leading to vocal cord paralysis and hypocalcemia. This study investigates whether topical application of methylene blue spray can enhance intraoperative visualization and preservation of these structures. A total of 136 patients with benign multinodular goiter were randomized into two groups: an experimental group receiving MB spray and a control group receiving conventional dissection. RLN injury was assessed via postoperative laryngoscopy, and serum calcium levels were measured at 72 hours postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* benign multinodular goiter scheduled for thyroidectomy.

Exclusion Criteria:

* Recurrent/metastatic disease
* Preoperative vocal cord dysfunction
* Coagulopathy
* Methylene blue allergy
* Hepatic/renal impairment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 136 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-01-20 (Actual)

PRIMARY OUTCOMES:
Incidence of recurrent laryngeal nerve injury | 2 hours (at extubation)
  Incidence of recurrent laryngeal nerve injury (assessed by indirect laryngoscopy
Postoperative serum calcium levels | At 72 hours
  Postoperative serum calcium levels

CONTACTS AND LOCATIONS:
Overall Officials: Awais Amjad Malik, MBBS, FCPS, Principal Investigator — Services Institute of Medical Sciences
Locations (1):
- Services Institute of Medical Sciences, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 6. Farghaly AEA, Ahmed MT, Kotb MB, Ibrahim IA. Conventional surgical techniques versus intraoperative methylene blue spraying for safe total thyroidectomy. J Curr Med Res Pract. 2019;4(1):67-71.
- [Background] 7. Sebaey AE, Khalil AM, Elkilany MM, Ali RM. Recurrent laryngeal nerve identification in thyroidectomy by intraoperative staining with methylene blue. Eur J Mol Clin Med. 2021;8(2):644-9.
- [Background] 8. Piromchai P, Juengtrakool T, Laohasiriwong S, Kasemsiri P, Ungarereevittaya P. The sensitivity and specificity of methylene blue spray to identify the parathyroid gland during thyroidectomy. PeerJ. 2019;7:e6376.
- [Background] 1. Eldeen Abdulrahman ZN, Rajab WQ, Jameel Ali Z. Identification of recurrent laryngeal nerve and parathyroid glands intraoperatively by methylene blue spraying technique. Indian J Forensic Med Toxicol. 2020;14(1):1355-60.